CLINICAL TRIAL: NCT01279044
Title: Reducing HIV Risk Among Episodic Substance Using Men Who Have Sex With Men (SUMSM): Adaptation of the Personalized Cognitive Counseling (PCC) Intervention
Brief Title: Reducing HIV Risk Among Episodic Substance Using Men Who Have Sex With Men (SUMSM)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: San Francisco Department of Public Health (Other Government)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Phillip Coffin, MD, MIA, Director of Substance Use Research, HIV Prevention, San Francisco Department of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1UR6PS000684-01 (NIH)
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infections; Episodic Substance Use
Keywords: HIV; MSM; SUMSM
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): HIV testing with adapted Personalized Cognitive Risk-reduction Counseling intervention (PCC)
  Interventions: Behavioral: Adapted Personalized Cognitive Risk-reduction Counseling intervention (PCC)
- 2 (Placebo Comparator): HIV testing with information only
  Interventions: Behavioral: Standard HIV testing with information only

INTERVENTIONS:
Behavioral: Adapted Personalized Cognitive Risk-reduction Counseling intervention (PCC) — The individualized, cognitive counseling intervention was designed to help participants address the self-justifications-beliefs, thoughts, and attitudes-that they employed in the setting of high-risk sexual behavior, in the company of an empathic counselor.
  Arms: 1
Behavioral: Standard HIV testing with information only — Standard HIV testing with information only
  Arms: 2

SUMMARY:
The purpose of this study is to determine if persons randomized to receive adapted Personalized Cognitive Risk-reduction Counseling (PCC) will report greater reductions in unprotected anal sex behavior compared with persons who do not receive Personalized Cognitive Risk-reduction Counseling (PCC).

DETAILED DESCRIPTION:
In the U.S., men who have sex with men (MSM) continue to constitute the greatest number of HIV/AIDS cases compared with other risk groups. Furthermore, many episodic substance using men who have sex with men (SUMSM) report that sex and substance use "always" or "often" go together. Studies have shown that substance use just before or during sex substantially increases HIV risk.

The formative phase of this research enrolled 59 HIV-negative episodic substance using MSM to participate in interviews to inform the adaptation of the Self-Justification Elicitation Instrument (SJEI) used during Personalized Cognitive Counseling (PCC) and to subsequently, pilot the adapted SJEI.

The randomized controlled trial (RCT) phase of this study enrolled 326 ethnically-diverse, HIV-negative episodic SUMSM to receive standard HIV rapid testing plus adapted Personalized Cognitive Risk-reduction Counseling intervention (PCC) or standard HIV counseling and rapid testing only.

Specific Aims:

1. To conduct formative research through individual interviews and pilot testing among a sample (n=59) of episodic substance-using men who have sex with men (SUMSM) to develop and adapt the key elements of the Personal Risk-Reduction Cognitive Counseling intervention, with a focus on eliciting and intervening on the thoughts, attitudes, and behaviors that episodic SUMSM employ when using substances and engaging in concurrent sexual risk.
2. To determine the efficacy of the adapted intervention in reducing unprotected anal sex, as compared to routine HIV testing control condition, in a randomized trial of 326 episodic SUMSM.

We will also determine the efficacy of the intervention in reducing substance use.

ELIGIBILITY:
Inclusion Criteria:

1. Reports within the past 6 months unprotected anal intercourse (UAI) with another man while under the influence of at least one or any combination of the following substance: methamphetamine, poppers, crack or powder cocaine, or alcohol if binge drinking (5 or more drinks) within 2 hours before or during sex.
2. Identifies as male.
3. HIV-negative or unknown serostatus by self-report
4. Willing and able to participate in an intervention that addresses episodic substance use and sexual risk behavior
5. Not currently in substance use treatment, a self-help program, or an HIV prevention study
6. Has not injected any substances in prior 6 months.
7. ≥ 18 years old
8. Planning to remain in the San Francisco Bay Area for the duration of study activities
9. Willing and able to provide full informed consent. Able to speak, read, and understand English.

Exclusion Criteria:

1. Reports within the past 6 months UAI with only one partner AND identifies that individual as a primary partner.
2. In the prior three months, weekly or more use of any of the targeted substances (meth, poppers, crack or powder cocaine), with the exception of alcohol
3. For alcohol, more than an average of 3 alcoholic drinks daily, or binge drinking more than twice weekly.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2007-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip O Coffin, MD, MIA, Principal Investigator — Director of Substance Use Research, HIV Prevention, San Francisco Department of Public Health; Jeffrey H Herbst, PhD, Study Director — Centers for Disease Control and Prevention
Locations (1):
- San Francisco Department of Public Health, AIDS Office, San Francisco, California, United States

REFERENCES:
- [Background] Santos GM, Coffin PO, Das M, Matheson T, DeMicco E, Raiford JL, Vittinghoff E, Dilley JW, Colfax G, Herbst JH. Dose-response associations between number and frequency of substance use and high-risk sexual behaviors among HIV-negative substance-using men who have sex with men (SUMSM) in San Francisco. J Acquir Immune Defic Syndr. 2013 Aug 1;63(4):540-4. doi: 10.1097/QAI.0b013e318293f10b. PMID 23572012
- [Background] Knight KR, Das M, DeMicco E, Raiford JL, Matheson T, Shook A, Antunez E, Santos GM, Dadasovich R, Dilley JW, Colfax GN, Herbst JH. A roadmap for adapting an evidence-based HIV prevention intervention: personal cognitive counseling (PCC) for episodic substance-using men who have sex with men. Prev Sci. 2014 Jun;15(3):364-75. doi: 10.1007/s11121-013-0364-z. PMID 23412947
- [Result] Coffin PO, Santos GM, Colfax G, Das M, Matheson T, DeMicco E, Dilley J, Vittinghoff E, Raiford JL, Carry M, Herbst JH. Adapted personalized cognitive counseling for episodic substance-using men who have sex with men: a randomized controlled trial. AIDS Behav. 2014 Jul;18(7):1390-400. doi: 10.1007/s10461-014-0712-4. PMID 24510401

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment involved outreach at community venues in San Francisco, including bars, clubs, grocery stores, gyms, and other venues frequented by MSM. To recruit a racially and ethnically diverse sample of episodic SUMSM, recruitment also occurred at community-based organizations serving African American, Latino, and Asian and Pacific Islander MSM.
Pre-assignment Details: Potential participants completed brief telephone screening to assess initial eligibility and, if eligible, were scheduled for in-person re-screening visits. If potential participants were ineligible at the re-screening visit, they were thanked for their time and did not continue with study activities, such as randomization in the RCT.
Groups:
- Formative Phase 1: Individual interviews and pilot testing to develop and adapt key elements of Personal Cognitive Counseling
- HIV Testing With Adapted Personalized Cognitive Risk-reduction: Adapted Personalized Cognitive Risk-reduction Counseling intervention (PCC): The individualized, cognitive counseling intervention was designed to help participants address the self-justifications-beliefs, thoughts, and attitudes-that they employed in the setting of high-risk sexual behavior, in the company of an empathic counselor.
- HIV Testing With Information Only: Standard HIV testing with information only: Standard HIV testing with information only
Period: PHASE 1 - Formative
Arm/Group | Formative Phase 1 | HIV Testing With Adapted Personalized Cognitive Risk-reduction | HIV Testing With Information Only
Started | 59 | 0 (Participants who participated in the formative phase did not participate in the RCT.) | 0 (Participants who participated in the formative phase did not participate in the RCT.)
Completed | 59 | 0 (Participants who participated in the formative phase did not participate in the RCT.) | 0 (Participants who participated in the formative phase did not participate in the RCT.)
Not Completed | 0 | 0 | 0
Period: PHASE 2 - Randmonized Controlled Trial
Arm/Group | Formative Phase 1 | HIV Testing With Adapted Personalized Cognitive Risk-reduction | HIV Testing With Information Only
Started | 0 (Participants who participated in the RCT did not participate in the formative phase.) | 162 | 164
Completed | 0 (Participants who participated in the RCT did not participate in the formative phase.) | 151 | 161
Not Completed | 0 | 11 | 3
Not completed — Withdrawal by Subject | 0 | 3 | 2
Not completed — Lost to Follow-up | 0 | 8 | 0
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: There were no significant differences between the two study arms on baseline demographics, HIV testing, and substance use. The mean age was 33.6 years; 49% were white and 51% non-white including 26% Latino/Hispanic, 11% Asian and Pacific Islander, 10% black/African American, and 6% mixed/other race.
Groups:
- Phase 1 - Formative Research: Formative research through individual interviews and pilot testing to develop and adapt the key elements of Personal Cognitive Counseling
- Total: Total of all reporting groups
Arm/Group | Phase 1 - Formative Research | HIV Testing With Adapted Personalized Cognitive Risk-reduction | HIV Testing With Information Only | Total
Number analyzed (Participants) | 59 | 162 | 164 | 385
Age, Continuous [Mean (Full Range); unit: years] | 33 [18 to 50] | 34 [18 to 61] | 33.1 [19 to 63] | 33.6 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 59 | 162 | 164 | 385
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 34 | 45 | 97
  Not Hispanic or Latino | 41 | 128 | 119 | 288
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black/African American | 3 | 17 | 16 | 36
  Asian Pacific Islander | 6 | 14 | 22 | 42
  Mixed | 3 | 12 | 12 | 27
  Native American | 1 | 1 | 1 | 3
  Other | 0 | 34 | 39 | 73
  White | 46 | 84 | 74 | 204
Region of Enrollment [Number; unit: participants]
  United States | 59 | 162 | 164 | 385

OUTCOME MEASURES:

1. Primary Outcome: Total Unprotected Anal Intercourse Events (Exclusive of Those Events With a Primary HIV-negative Partner)
Description: The outcome measure data shows the rate of change in the mean value in the number of total unprotected anal intercourse events over time. Behaviors were self-reported at each study visit using "during the past 3 months" as the recall period. Study visits took place at baseline, 3 month, and 6 month timepoints.
Time Frame: Self-reported behavior during past 3 months
Measure: Number; unit: Self reported events in past 3 months
Arm/Group | HIV Testing With Adapted Personalized Cognitive Risk-reduction | HIV Testing With Information Only
Number analyzed (Participants) | 162 | 164
Self reported events in past 3 months
  Mean number at baseline | 4.23 | 3.91
  Mean number at 3 months | 3.41 | 2.05
  Mean number at 6 months | 1.83 | 1.96
  Rate of change in mean value of outcome over time | 0.47 | 0.45

2. Primary Outcome: Total Unprotected Anal Intercourse Partners
Description: The outcome measure data shows the rate of change in the mean value of total unprotected anal intercourse partners over time. Behaviors were self-reported at each study visit using "during the past 3 months" as the recall period. Study visits took place at baseline, 3 month, and 6 month timepoints.
Time Frame: Self-reported behavior during past 3 months
Measure: Number; unit: Partners in past 3 months
Arm/Group | HIV Testing With Adapted Personalized Cognitive Risk-reduction | HIV Testing With Information Only
Number analyzed (Participants) | 162 | 164
Partners in past 3 months
  Mean number of partners at baseline | 2.71 | 2.60
  Mean number of partners at 3 months | 1.54 | 1.37
  Mean number of partners at 6 months | 1.27 | 1.16
  Rate of change in mean value of outcome over time | 0.46 | 0.43

3. Primary Outcome: Unprotected Anal Intercourse Episodes With Three Most Recent Sex Partners at Each Follow-up Visit, Exclusive of Primary HIV-negative Partners.
Description: The outcome measure data shows the rate of change in the mean value of total unprotected anal intercourse episodes with three most recent sex partners over time. Behaviors were self-reported at each study visit using "during the past 3 months" as the recall period. Study visits took place at baseline, 3 month, and 6 month timepoints.
Time Frame: Self-reported behavior during past 3 months
Measure: Number; unit: Episodes in past 3 months
Arm/Group | HIV Testing With Adapted Personalized Cognitive Risk-reduction | HIV Testing With Information Only
Number analyzed (Participants) | 162 | 164
Episodes in past 3 months
  Mean number of episodes at baseline | 1.97 | 2.31
  Mean number of episodes at 3 months | 1.12 | 1.11
  Mean number of episodes at 6 months | 0.83 | 1.20
  Rate of change in mean value of outcome over time | 0.39 | 0.52

4. Secondary Outcome: Number of Serodiscordant Unprotected Anal Intercourse (SDUAI) Events
Description: The outcome measure data shows the rate of change in the mean value of number of serodiscordant unprotected anal intercourse events. Behaviors were self-reported at each study visit using "during the past 3 months" as the recall period. Study visits took place at baseline, 3 month, and 6 month timepoints.
  Serodiscordant defined as having partner of discordant or of unknown HIV serostatus.
Time Frame: Self-reported behavior during past 3 months
Measure: Number; unit: Events in past 3 months
Arm/Group | HIV Testing With Adapted Personalized Cognitive Risk-reduction | HIV Testing With Information Only
Number analyzed (Participants) | 162 | 164
Events in past 3 months
  Mean number of events at baseline | 1.06 | 1.13
  Mean number of events at 3 months | 0.43 | 0.49
  Mean number of events at 6 months | 0.34 | 0.55
  Rate of change in mean value of outcome over time | 0.28 | 0.47

5. Secondary Outcome: Number of Instertive UAI Events
Description: The outcome measure data shows the rate of change in the mean value of number of instertive unprotected anal intercourse (UAI) events. Behaviors were self-reported at each study visit using "during the past 3 months" as the recall period. Study visits took place at baseline, 3 month, and 6 month timepoints.
Time Frame: Self-reported behavior during past 3 months
Measure: Number; unit: Self reported behavior in past 3 months
Arm/Group | HIV Testing With Adapted Personalized Cognitive Risk-reduction | HIV Testing With Information Only
Number analyzed (Participants) | 162 | 164
Self reported behavior in past 3 months
  Mean number of events at baseline | 2.84 | 2.44
  Mean number of events at 3 months | 2.80 | 1.32
  Mean number of events at 6 months | 1.37 | 1.14
  Rate of change in mean value over time | 0.55 | 0.41

6. Secondary Outcome: Number of Receptive UAI Events
Description: The outcome measure data shows the rate of change in the mean value of the number of receptive unprotected anal intercourse (UAI) events. Behaviors were self-reported at each study visit using "during the past 3 months" as the recall period. Study visits took place at baseline, 3 month, and 6 month timepoints.
Time Frame: Self-reported behavior during past 3 months
Measure: Number; unit: Self reported behavior in past 3 months
Arm/Group | HIV Testing With Adapted Personalized Cognitive Risk-reduction | HIV Testing With Information Only
Number analyzed (Participants) | 162 | 164
Self reported behavior in past 3 months
  Mean number of events at baseline | 1.39 | 1.48
  Mean number of events at 3 months | 0.61 | 0.73
  Mean number of events at 6 months | 0.45 | 0.82
  Rate of change in mean value of outcome over time | 0.31 | 0.53

7. Secondary Outcome: Number of Condom-protected Anal Intercourse Events
Description: The outcome measure data shows the rate of change in the mean value of the number of condom-protected anal intercourse (UAI) events. Behaviors were self-reported at each study visit using "during the past 3 months" as the recall period. Study visits took place at baseline, 3 month, and 6 month timepoints.
  Serodiscordant defined as having partner of discordant or of unknown HIV serostatus.
Time Frame: Self-reported behavior during past 3 months
Measure: Number; unit: Self reported behavior in past 3 months
Arm/Group | HIV Testing With Adapted Personalized Cognitive Risk-reduction | HIV Testing With Information Only
Number analyzed (Participants) | 162 | 164
Self reported behavior in past 3 months
  Mean number of events at baseline | 3.78 | 2.83
  Mean number of events at 3 months | 1.67 | 2.13
  Mean number of events at 6 months | 2.11 | 1.29
  Rate of change in mean value of outcome over time | 0.57 | 0.44

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | HIV Testing With Adapted Personalized Cognitive Risk-reduction | HIV Testing With Information Only
Serious Adverse Events (participants affected / at risk) | 0/162 | 1/164
Other Adverse Events (participants affected / at risk) | 0/162 | 0/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV Testing With Adapted Personalized Cognitive Risk-reduction (N=162) | HIV Testing With Information Only (N=164)
Death (Psychiatric disorders) | 0 | 1 (1) — Suicide

LIMITATIONS AND CAVEATS:
Self-report data subject to recall bias Sample is San Francisco SUMSM; may not be generalizable to other locations 42% screened as substance-dependent per SDS Inclusion of dependent MSM reduced ability to detect significant intervention effects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No